CLINICAL TRIAL: NCT03848910
Title: Subject´s Preference Regarding Hearing Performance and Functionality Using a New Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5731
Record Dates: First submitted 2019-02-08; First posted 2019-02-21 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-01

CONDITIONS: Deafness; Sensoneural Single Sided; Conductive Hearing Loss; Mixed Hearing Loss
MeSH Terms: conditions — Deafness; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational device - Sound Processor (Experimental)
  Interventions: Device: Investigational device - Sound Processor

INTERVENTIONS:
Device: Investigational device - Sound Processor — At visit 1 the subjects will complete self-reported assessments with respect to "pre-study experience" using precursor Sound Processor (comparator). At visit 1 the subjects will then receive the Investigational device (Sound Processor) which should be used during the following 6 weeks. At visit 3 the subjects will complete self-reported assessments regarding Investigational device and participate in audiology tests regarding both Sound Processors, comparator and Investigational device. The subject shall decide their preferred choice made by selection between Investigational device and the comparator.

SUMMARY:
The aim of this clinical investigation is to investigate the subject´s overall preference, hearing performance and self-reported assessments with the Investigational device and its precursor Sound Processor (Comparator) after 6 weeks in subjects with conductive/mixed hearing loss or Single Sided Deafness, (SSD).

ELIGIBILITY:
Inclusion Criteria:

* Completed clinical investigation CBAS5539, and an active user of the Osia System.
* Signed Informed consent.
* Subject with conductive or mixed hearing loss in the implanted ear. Bone conduction thresholds with pure tone average (PTA4; mean of 0.5, 1, 2 and 4 kHz) of ≤ 55 dB HL.

OR subject with single-sided sensorineural deafness. Air conduction thresholds with a pure tone average PTA4 of ≤ 20 dB (decibel) HL (Hearing Level) (mean of 0.5, 1, 2 and 3 kHz) in the good ear.

- Optimally fitted with Osia Sound processor, according to subject's experience prior to inclusion.

Exclusion Criteria:

* Any ongoing soft tissue complication that could significantly affect the use of the Osia 2 Sound Processor during the 6 weeks period
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator
* Unable to follow investigational procedures and instructions, e.g. inability to complete quality of life scales or audiological testing as described in the Clinical Investigation Plan (CIP).
* Participation in another clinical investigation with pharmaceutical and/or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cowan, Prof, Principal Investigator — HEARing CRC550, Carlton, Melbourne
Locations (1):
- HEARing CRC550 Swanston Street, Carlton, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device - Sound Processor
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Investigational Device - Sound Processor: Investigational device - Sound Processor: At visit 1 the subjects completed self-reported assessments with respect to "pre-study experience" using precursor Sound Processor (comparator). At visit 1 the subjects then received the Investigational device (Sound Processor) which was used during the following 6 weeks. At visit 3 the subjects completed self-reported assessments regarding Investigational device and participated in audiology tests regarding both Sound Processors, comparator and Investigational device. The subject decided their preferred choice made by selection between Investigational device and the comparator.
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Australia | 11

OUTCOME MEASURES:

1. Primary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: Measuring of subscales Ease of communication, Reverberation, Background noise, Aversiveness and a Global score with the precursor sound processor at Day 0 and with the Investigational device after 6 weeks with a questionnaire. All subscales range from 0-100%, total score is the average of all subscales 0-100%, where 0% indicates no problems and 100% indicates always problem. A decrease in the APHAB values indicates an improvement. The change from visit 1 with the precursor sound processor to visit 3 with the Investigational device is presented. A positive value indicates an improvement with the Investigational device, a negative value an impairment.
Time Frame: Day 0 (Visit 1) and after 6 weeks (Visit 3)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
units on a scale
  Ease of communication | 6.3 (10.1)
  Background noise | 7.0 (12.6)
  Reverberation | 5.6 (10.3)
  Aversiveness | 3.5 (7.5)
  Global | 6.3 (9.5)

2. Primary Outcome: Speech, Spatial, and Qualities of Hearing Scale (SSQ)
Description: Measuring speech, spatial and hearing experiences with the precursor sound processor at Day 0 (Visit 1) and with Investigational device after 6 weeks (Visit 3) with a questionnaire. The Total score summarizes the parameters speech, spatial and hearing. A scale from 0 to 10, where 0 represents "can not hear at all", and 10 "hear perfectly" is used. An increase of a SSQ value reflects an improvement. The change from visit 1 with the precursor sound processor to visit 3 with the Investigational device is presented. A positive value indicates an improvement and a negative value an impairment.
Time Frame: Day 0 and after 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
units on a scale
  Spatial score | 1.0 (1.6)
  Quality score | 0.061 (1.26)
  Speech | 0.96 (0.89)
  Total | 0.68 (0.62)

3. Primary Outcome: Self-reported Assessment Regarding Satisfaction and Usability (QUEST Version 2)
Description: Measuring QUEST (Self-reported assessment regarding satisfaction and usability) using a questionnaire, with the precursor sound processor at Day 0 (Visit 1) and with the Investigational device after 6 weeks (Visit 3). The QUEST form displays the scoring of 8 satisfaction items. The satisfaction items related to the characteristics of the device are: 1) dimensions, 2) weight, 3) adjustments, 4) safety, 5) durability, 6) simplicity of use, 7) comfort and 8) effectiveness. A scale from 1 to 5, where 1 represent not satisfied at all, 2 not very satisfied, 3 more or less satisfied, 4 quiet satisfied and 5 represents very satisfied.
  The three most important items of 1) dimensions, 2) weight, 3) adjustments, 4) safety, 5) durability, 6) simplicity of use, 7) comfort and 8) effectiveness were listed by each participant.
Time Frame: Day 0 and after 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Visit 1: Dimension; not satisfied at all | 0
  Visit 1: Dimension; not very satisfied | 0
  Visit 1: Dimension; more or less satisfied | 3
  Visit 1: Dimension; quiet satisfied | 4
  Visit 1: Dimension; very satisfied | 4
  Visit 3: Dimension; not satisfied at all | 0
  Visit 3: Dimension; not very satisfied | 0
  Visit 3: Dimension; more or less satisfied | 0
  Visit 3: Dimension; quiet satisfied | 3
  Visit 3: Dimension; very satisfied | 8
  Visit 1: Weight; not satisfied at all | 0
  Visit 1: Weight; not very satisfied | 0
  Visit 1: Weight; more or less satisfied | 0
  Visit 1: Weight; quiet satisfied | 3
  Visit 1: Weight; very satisfied | 8
  Visit 3: Weight; not satisfied at all | 0
  Visit 3: Weight; not very satisfied | 0
  Visit 3: Weight; more or less satisfied | 0
  Visit 3: Weight; quiet satisfied | 0
  Visit 3: Weight; very satisfied | 11
  Visit 1: Adjustment; not satisfied at all | 0
  Visit 1: Adjustment; not very satisfied | 0
  Visit 1: Adjustment; more or less satisfied | 2
  Visit 1: Adjustment; quiet satisfied | 3
  Visit 1: Adjustment; very satisfied | 6
  Visit 3: Adjustment; not satisfied at all | 0
  Visit 3: Adjustment; not very satisfied | 0
  Visit 3: Adjustment; more or less satisfied | 1
  Visit 3: Adjustment; quiet satisfied | 2
  Visit 3: Adjustment; very satisfied | 8
  Visit 1: Safety; not satisfied at all | 0
  Visit 1: Safety; not very satisfied | 0
  Visit 1: Safety; more or less satisfied | 3
  Visit 1: Safety; quiet satisfied | 1
  Visit 1: Safety; very satisfied | 7
  Visit 3: Safety; not satisfied at all | 0
  Visit 3: Safety; not very satisfied | 1
  Visit 3: Safety; more or less satisfied | 2
  Visit 3: Safety; quiet satisfied | 2
  Visit 3: Safety; very satisfied | 6
  Visit 1: Durability; not satisfied at all | 0
  Visit 1: Durability; not very satisfied | 0
  Visit 1: Durability; more or less satisfied | 1
  Visit 1: Durability; quiet satisfied | 4
  Visit 1: Durability; very satisfied | 6
  Visit 3: Durability; not satisfied at all | 0
  Visit 3: Durability; not very satisfied | 0
  Visit 3: Durability; more or less satisfied | 1
  Visit 3: Durability; quiet satisfied | 4
  Visit 3: Durability; very satisfied | 6
  Visit 1: Easy of use; not satisfied at all | 0
  Visit 1: Easy of use; not very satisfied | 0
  Visit 1: Easy of use; more or less satisfied | 3
  Visit 1: Easy of use; quiet satisfied | 3
  Visit 1: Easy of use; very satisfied all | 5
  Visit 3: Easy of use; not satisfied at all | 0
  Visit 3: Easy of use; not very satisfied | 0
  Visit 3: Easy of use; more or less satisfied | 1
  Visit 3: Easy of use; quiet satisfied | 3
  Visit 3: Easy of use; very satisfied all | 7
  Visit 1: Comfort; not satisfied at all | 0
  Visit 1: Comfort; not very satisfied | 0
  Visit 1: Comfort; more or less satisfied | 0
  Visit 1: Comfort; quiet satisfied | 3
  Visit 1: Comfort; very satisfied | 8
  Visit 3: Comfort; not satisfied at all | 0
  Visit 3: Comfort; not very satisfied | 0
  Visit 3: Comfort; more or less satisfied | 0
  Visit 3: Comfort; quiet satisfied | 2
  Visit 3: Comfort; very satisfied | 9
  Visit 1: Effectiveness; not satisfied at all | 0
  Visit 1: Effectiveness; not very satisfied | 0
  Visit 1: Effectiveness; more or less satisfied | 1
  Visit 1: Effectiveness; quiet satisfied | 7
  Visit 1: Effectiveness; very satisfied | 3
  Visit 3: Effectiveness; not satisfied at all | 0
  Visit 3: Effectiveness; not very satisfied | 0
  Visit 3: Effectiveness; more or less satisfied | 1
  Visit 3: Effectiveness; quiet satisfied | 3
  Visit 3: Effectiveness; very satisfied | 7
  Visit 1: Important item, Dimensions | 2
  Visit 1: Important item, Weight | 1
  Visit 1: Important item, Adjustments | 2
  Visit 1: Important item, Safety | 0
  Visit 1: Important item, Durability | 5
  Visit 1: Important item, Easy of use | 5
  Visit 1: Important item, Comfort | 7
  Visit 1: Important item, Effectiveness | 11
  Visit 3: Important item, Dimensions | 4
  Visit 3: Important item, Weight | 0
  Visit 3: Important item, Adjustments | 1
  Visit 3: Important item, Safety | 1
  Visit 3: Important item, Durability | 5
  Visit 3: Important item, Easy of use | 4
  Visit 3: Important item, Comfort | 7
  Visit 3: Important item, Effectiveness | 11

4. Primary Outcome: Audiometric Thresholds in Freefield, Pure Tone Average 4 (PTA4)
Description: To measure threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz) with both the precursor sound processor and the Investigational device. The units reported for PTA4 are decibels (dB). The change from visit 1 with the precursor sound processor to visit 3 with the Investigational device is presented. As such, a lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: Baseline at visit 1, 6 weeks after study start at visit 3
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
dB | -2.5 (2.4)

5. Primary Outcome: Audiometric Thresholds in Freefield, Individual Frequencies
Description: To measure threshold audiometry at individual frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 Hz with both the precursor sound processor and the Investigational device. The units reported for threshold audiometry are decibels (dB). The change from visit 1 with the precursor sound processor to visit 3 with the Investigational device is presented. As such, a lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: 6 weeks after study start
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
dB
  250 Hz | -2.3 (4.7)
  500 Hz | -3.6 (5.1)
  750 Hz | -6.4 (3.9)
  1000 Hz | -3.6 (3.9)
  1500 Hz | -3.6 (6.0)
  2000 Hz | -1.2 (3.4)
  3000 Hz | -4.1 (3.8)
  4000 Hz | -0.9 (5.4)
  6000 Hz | -4.6 (4.2)
  8000 Hz | -1.8 (14.7)

6. Primary Outcome: Adaptive Speech Recognition in Noise Ratio
Description: To measure Adaptive speech recognition in noise with the precursor sound processor and the Investigational device. Measured as signal to noise ratio The adaptive speech test in noise was conducted using validated lists of phonetically balanced sentences, with speech and noise presented from the front (0 degrees azimuth). The speech is kept constant at 65 dB Sound Pressure Level (SPL) and the noise is adapted in dB steps to establish the speech-to-noise ratio (SNR) providing a 50% level of understanding. A ratio of 1 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A lower ratio than 1 reflects the ability to correctly hear sentences below 65 dB. A ratio higher than 1 reflects the ability to correctly hear sentences presented above 65 dB. A lower or more negative score is more desirable and represent a better hearing in a noisy environment.
Time Frame: Baseline at visit 1, 6 weeks after study start at visit 3
Measure: Mean (Standard Deviation); unit: SNR
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
SNR
  Visit 1 | -1.3 (1.2)
  Visit 3 | -1.2 (1.4)

7. Primary Outcome: Speech in Quiet
Description: To measure Speech in quiet at 50, 65 and 80 dB with the precursor sound processor and the Investigational device. Speech in Quiet presents a list of words in a quiet environment at three different presentations levels, 50, 65 and 80 dB (decibel). The number of correct words perceived at each presentation level are counted and the percentage in relation to the total presented amount of words is calculated. A higher score reflects a higher percentage of correct words perceived, i.e. better hearing in a quiet environment.
Time Frame: Baseline at visit 1, 6 weeks after study start at visit 3
Measure: Mean (Standard Deviation); unit: % correct perceived words
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
% correct perceived words
  50 dB visit 1 | 82.5 (6.8)
  50 dB visit 3 | 83.3 (7.2)
  65 dB visit 1 | 93.7 (2.4)
  65 dB visit 3 | 96.9 (2.4)
  80 dB visit 1 | 94.4 (4.1)
  80 dB visit 3 | 96.9 (2.6)

8. Primary Outcome: To Compare the Subject´s Overall Preference Regarding the Investigational Device and the Precursor Sound Processor
Description: The test subject will be asked a question regarding preferred choice made by selection between Investigational device and the precursor sound processor (comparator). Three boxes can be ticked; Precursor Sound Processor, Investigational Device, No preference.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  No preference | 0
  Precursor sound processor | 0
  Investigational device | 11

9. Primary Outcome: To Assess the Subject's Experience Regarding Comfort
Description: Measure Comfort by a visual analogue scale (VAS) 100 mm at Day 0 regarding the precursor sound processor and after 6 weeks regarding the Investigational device. Subject will be asked to put a line where they find most appropriate where 0 mm represents Not comfortable at all and 100 represents Most comfortable imaginable. The distance will be measured with a ruler and presented as a value between 0 and 100. A higher score reflects higher comfort.
Time Frame: Baseline at visit 1, 6 weeks after study start at visit 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
units on a scale
  Precursor sound processor | 84.9 (16.8)
  Investigational device | 87.5 (7.5)

10. Primary Outcome: To Assess the Subject's Experience Regarding Usage; Magnet Choice
Description: Magnet choice will be entered; four boxes are available, 1, 2, 3 and 4, the box with the strength chosen by the patient will be ticked. Magnet strength 1 is the weakest and 4 is the strongest.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Strength 1 | 1
  Strength 2 | 3
  Strength 3 | 3
  Strength 4 | 4

11. Primary Outcome: To Assess the Subject's Experience Regarding Usage; Battery Life Time
Description: The patient will be asked a question regarding battery life; "How often was the battery changed". A free text field is available for answer.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Every day | 2
  Two work days (16 hours) | 1
  1.5 days | 2
  Every 2 days | 3
  Every 3 days | 1
  Every 3-4 days | 1
  1-2 times a week | 1

12. Primary Outcome: To Assess the Subject's Experience Regarding Usage; Softwear Pad
Description: The patient will be asked a question "Did you use a SoftWear Pad in the last 6 weeks". The patient can tick a "Yes" or "No" box.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Yes | 2
  No | 9

13. Primary Outcome: To Assess the Subject's Experience Regarding Usage; Safety Line
Description: The patient will be asked a question "Did you use a safety line in the last 6 weeks". The patient can tick a "Yes" or "No" box.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Yes | 9
  No | 2

14. Primary Outcome: To Assess the Subject's Experience Regarding Usage; Wireless Accessories
Description: The patient will be asked a question "Did you use a Wireless accessory during the last 6 weeks". The patient can tick a "Yes" or "No" box.
Time Frame: 6 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device - Sound Processor
Number analyzed (Participants) | 11
Participants
  Yes | 11
  No | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Investigational Device - Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device - Sound Processor (N=11)
Skin irritation-test ear (Skin and subcutaneous tissue disorders) | 1 (1)
Fluid in middle ear (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Mastoid cavity infection (Infections and infestations) | 1 (1)
Fall due to SCCD (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution must give a copy of any proposed Publication to the Sponsor at least 40 days before forwarding it to any person that is not bound by the confidentiality obligations

The Sponsor may, within that 40-day period:

1. provide comments;
2. request delay of Publication for no more than 120 days, or
3. request that the Discloser remove specified Confidential Information from the Publication.

DOCUMENTS (2):
  • Study Protocol (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT03848910/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT03848910/SAP_000.pdf